CLINICAL TRIAL: NCT05664958
Title: Erector Spinae Plane Block With Liposomal Bupivacaine for Post Cesarean Delivery Analgesia: A Pilot Study
Brief Title: ESP Block for Post Cesarean Analgesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00112152
Record Dates: First submitted 2022-12-09; First posted 2022-12-27 (Actual); Results first posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Cesarean Section Complications
MeSH Terms: interventions — Parapsychology; Dental Occlusion; Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- ESP Block (Experimental): Standard of care analgesic regimen with ESP Block
  Interventions: Procedure: Erector Spinae Plane (ESP) Block; Drug: bupivacaine liposome injectable suspension; Drug: bupivacaine
- Control (No Intervention): Standard of care analgesic regimen

INTERVENTIONS:
Procedure: Erector Spinae Plane (ESP) Block — ESP Block with liposomal bupivacaine and immediate release bupivacaine
  Arms: ESP Block
Drug: bupivacaine liposome injectable suspension — 133 mg liposomal bupivacaine per side.
  Arms: ESP Block
Drug: bupivacaine — 20 ml bupivacaine 0.25% per side.
  Arms: ESP Block

SUMMARY:
The purpose of this pilot study is to assess the analgesic efficacy of Erector Spinae Plane block (ESPB) with liposomal bupivacaine in women undergoing cesarean delivery and receiving a postoperative multimodal analgesic regimen as assessed by the dose of rescue postoperative opioids compared to a historical control group of women receiving the same multimodal regimen but with no truncal blocks. This will be a case control study with a prospective and a retrospective component. Women undergoing elective cesarean delivery under spinal or combined spinal epidural anesthesia will be approached to participate in the prospective open label component of the study. Cases will be matched in a 1:4 ratio by age, race, history of prior cesarean delivery, and insurance status with historical controls who received the same multimodal analgesic regimen but no truncal blocks. We plan to enroll 30 subjects for the prospective arm of the study and 120 for the retrospective arm.

DETAILED DESCRIPTION:
This will be a case control study with a prospective and a retrospective component. Women undergoing elective cesarean delivery under spinal or combined spinal epidural anesthesia will be approached to participate in the prospective open label component of the study. Those women will receive the standard of care intraoperative and postoperative analgesic regimen used at Duke university incorporating 100 mcg intrathecal morphine, intraoperative acetaminophen 975 mg PR and ketorolac 15 mg IV and postoperative scheduled oral acetaminophen 975 mg every 6 hours, scheduled 15 mg IV ketorolac for 3 doses every 6 hours followed by oral ibuprofen 600 mg every 6 hours. At the end of surgery, a bilateral ESPB will be performed under ultrasound guidance using 133 mg liposomal bupivacaine and 20 ml bupivacaine 0.25% per side.

Cases will be matched in a 1:4 ratio by age, race, history of prior cesarean delivery, and insurance status with historical controls who received the same multimodal analgesic regimen but no truncal blocks.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years of age with a term pregnancy of 37 to 42 weeks and American Society of Anesthesiologists Physical Status Classification II or III scheduled to undergo elective CD.

Exclusion Criteria:

* ≥3 prior CDs, pre-pregnancy body mass index >40 kg/m2, planned concurrent surgical procedure other than tubal ligation, chronic pain or chronic opioid therapy, any clinically significant event or condition uncovered during surgery (eg, excessive bleeding, acute sepsis) that might render the patient medically unstable or complicate the patient's postsurgical course, or allergy or contraindication to any component of the multimodal analgesic regimen.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2023-04-17 (Actual); Primary Completion 2023-11-09 (Actual); Study Completion 2023-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf S Habib, MD, Principal Investigator — Duke University Hospital
Locations (1):
- Duke University Hospital, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Feldman S, Holmes RJ Jr, Fuller M, Habib AS. Erector spinae plane block with liposomal bupivacaine for post-cesarean analgesia. Int J Gynaecol Obstet. 2025 Jul;170(1):489-495. doi: 10.1002/ijgo.70027. Epub 2025 Feb 21. PMID 39981694

RESULTS

PARTICIPANT FLOW:
Groups:
- Historical Control: Standard of care analgesic regimen
Period: Overall Study
Arm/Group | ESP Block | Historical Control
Started | 30 | 120
Completed | 30 | 120
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ESP Block | Historical Control | Total
Number analyzed (Participants) | 30 | 120 | 150
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 120 | 150
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 33 [29 to 36] | 33 [30 to 36] | 33 [29 to 36]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 120 | 150
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 16 | 20
  White | 23 | 92 | 115
  More than one race | 1 | 4 | 5
  Unknown or Not Reported | 2 | 8 | 10
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 120 | 150

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Oxycodone Consumption 0- 48 Hours After Cesarean Delivery
Description: Total dose of rescue oxycodone used in mg 0- 48 hours after cesarean delivery
Time Frame: 0-48 hours after cesarean delivery
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | ESP Block | Historical Control
Number analyzed (Participants) | 30 | 120
mg | 12.5 [5 to 40] | 25 [3.8 to 50]

2. Secondary Outcome: Postoperative Opioid Consumption at 24 Hours
Description: Total dose of rescue opioids used in mg oral morphine equivalents (OME) at 24 hours after cesarean delivery. OME are approximations of the equianalgesic effects of other opioids compared to oral morphine. Thus, OMEs indicate how much of the reference drug oral morphine would be required to treat pain as effectively as the comparison opioid.
Time Frame: 0-24 hours
Measure: Median (Inter-Quartile Range); unit: mg OME
Arm/Group | ESP Block | Historical Control
Number analyzed (Participants) | 30 | 120
mg OME | 7.5 [0 to 22.5] | 15 [0 to 30]

3. Secondary Outcome: Time to First Postsurgical Opioid Rescue Medication
Description: Time to first rescue opioid medication used for the treatment of breakthrough pain
Time Frame: 0-48 hours
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | ESP Block | Historical Control
Number analyzed (Participants) | 30 | 120
hours | 12.2 [4.7 to 30.2] | 3.2 [1.7 to 13.1]

4. Secondary Outcome: Area Under the Curve (AUC) of Verbal Rating Scale (VRS) Pain Intensity Scores
Description: Area under the curve (AUC) of verbal rating scale (VRS) pain intensity scores, lower scores indicate a better outcome. The VRS consists of a scale of 0 ('no pain') to 10 ('pain as bad as it could possibly be').
Time Frame: 0-48 hours
Measure: Median (Inter-Quartile Range); unit: pain score unit*hours
Arm/Group | ESP Block | Historical Control
Number analyzed (Participants) | 30 | 120
pain score unit*hours | 115 [26 to 151] | 140 [86 to 180]

5. Secondary Outcome: Number of Participants With Postoperative Nausea and Vomiting
Description: Occurrence of nausea and vomiting 0-48 h after cesarean delivery
Time Frame: 0-48 hours
Population: Data about postoperative nausea and vomiting not collected on the control group.
Measure: Count of Participants; unit: Participants
Arm/Group | ESP Block | Historical Control
Number analyzed (Participants) | 30 | 0
Participants | 12 |

6. Secondary Outcome: Number of Participants With the Need for Rescue Antiemetics
Description: Number of participants who needed medications to treat nausea and vomiting
Time Frame: 0-48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | ESP Block | Historical Control
Number analyzed (Participants) | 30 | 120
Participants | 8 | 48

7. Secondary Outcome: Number of Participants With Pruritus
Description: Number of participants who complained of pruritus
Time Frame: 0-48 hours
Population: Data about pruritus not collected on the control group.
Measure: Count of Participants; unit: Participants
Arm/Group | ESP Block | Historical Control
Number analyzed (Participants) | 30 | 0
Participants | 21 |

8. Secondary Outcome: Number of Participants With the Need for Rescue Antipruritics
Description: Number of participants who needed medications for treatment for pruritus
Time Frame: 0-48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | ESP Block | Historical Control
Number analyzed (Participants) | 30 | 120
Participants | 5 | 30

9. Secondary Outcome: Number of Participants Not Receiving Any Rescue Opioids Postoperatively
Description: Number of participants who did not need any opioids for break through pain
Time Frame: 0-48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | ESP Block | Historical Control
Number analyzed (Participants) | 30 | 120
Participants | 6 | 27

ADVERSE EVENTS:
Time Frame: Up to 48 hours
Arm/Group | ESP Block | Control
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/120
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/120
Other Adverse Events (participants affected / at risk) | 0/30 | 0/120

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-10-01): https://cdn.clinicaltrials.gov/large-docs/58/NCT05664958/Prot_SAP_000.pdf